# **Title of Research Study:**

Transgender men's perspectives on HIV risk and HIV prevention interventions.

**Principal Investigator:** Ricky Hill, Ph.D.

**Document Date:** June 14<sup>th</sup>, 2022

## Title of Research Study:

Transgender men's perspectives on HIV risk and HIV prevention interventions.

Principal Investigator: Ricky Hill, Ph.D.

**Student Investigator:** N/A

**Supported By:** Pilot award from the Third Coast Center for AIDS Research (CFAR), an NIH-funded center (P30AI117943), with co-funding from the following Institutes and Centers: NICHD, NIA, NIDCR, NINR, NHLBI, NICHD, NIDA, NIDDK, NIMHD, NIMH, NCI, NIAID, FIC, and OAR.

#### **Conflict of Interest Disclosure:**

We have no conflicts of interest relevant to this study to disclose.

#### **Key Information about this research study:**

The following is a short summary to help you decide whether to join this study. You can find more detailed information later in this form.

- The **purpose of this study** is to gather information through focus groups with transgender men and transmasculine people who have sex with cisgender men to learn more about the intersections of gender and sexual identities. We also want to better understand how life experiences unique to transgender men and transmasculine people influence their attitudes and beliefs about HIV risk. Together, this information will be key in developing and tailoring effective HIV prevention interventions to the transmasculine community.
- You will complete an online demographic survey. You will also participate in one, two-hour long focus group with other transgender men and transmasculine people where you will be asked questions about 1) how you find sexual partners; 2) perceptions of HIV risk; 3) sexual behavior; 4) HIV prevention strategies; and 5) sexual health and HIV prevention information preferences.
- Your participation in this study will be done either remotely via Zoom video conferencing OR
  it will be done in person at our research lab in downtown Chicago, at 625 N Michigan Ave.
  You will be asked about your location preferences at time of study contact.
- The **primary potential risk** of participation is breach of confidentiality. For example, there is a small chance that others might get access to your self-reported information, such as your transgender status. Another potential risk is discomfort from sensitive questions.
- The **main benefit** of being in this study is helping researchers learn about the intersection of gender and sexual identities and how that influences attitudes and behaviors about HIV prevention and sexual health. You are helping guide the future of transgender health interventions by participating in this study.

### Why am I being asked to take part in this research study?

We are asking you to take part in this research study because you:

1. Identify as a transgender man or transmasculine person.

- 2. Are over 18 years old.
- 3. Have sex with/sexual attraction to cisgender men.
- 4. Agree to the audio recording of focus groups.

## How many people will be in this study?

We expect 30 people will be in this study.

### What should I know about participating in a research study?

- Our research staff will explain the research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.
- You do not have to answer any question you do not want to answer.

### What happens if I say, "Yes, I want to be in this research"?

You will first fill out an online questionnaire that asks about your demographics. Next, you will be contacted by someone from the study team to determine if an online or in-person focus group is best for you, and you will be scheduled for one of the two-hour long focus group sessions. This focus group will ask questions about 1) how you find sexual partners; 2) perceptions of HIV risk; 3) sexual behavior; 4) HIV prevention strategies; and 5) sexual health and HIV prevention information preferences.

All focus group sessions will be audio recorded so that we have detailed information on how to create tailored HIV prevention programs for transgender men and transmasculine people. Audio recording will be completed using an external audio recorder. While some sessions may take place over the videoconference platform Zoom, no audio or video recordings of any nature will be saved to Zoom. Agreeing to the audio recording is required for participation. If you do not wish to be recorded, you cannot participate in this study.

#### Will being in this study help me in any way?

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits include:

- 1. Learning from other transgender men and transmasculine people.
- 2. Sharing information and skills that might help other transgender men and transmasculine people improve their sexual health and HIV prevention strategies.
- 3. Helping scientists to learn about how to reduce HIV risks and health disparities among transgender men and transmasculine people who have sex with cisgender men. So, you being in this study could help transgender men and transmasculine people like you in the future.

## Is there any way being in this study could be bad for me?

A possible risk for any research is <u>breach of confidentiality</u>. This means that people outside the study might get hold of your study information. We will do everything we can to minimize this risk. You can find more details later in this form.

<u>Some questions might make you feel uncomfortable</u>. If this happens in the demographics survey, you can skip the question. If this happens during the focus group session, you can leave the discussion or not answer the question. You can also leave the study completely.

### What happens if I do not want to be in this research, or I change my mind later?

Participation in research is voluntary. You can decide to participate or not to participate. If you do not want to be in this study or withdraw from the study at any point, simply tell our staff about it. Your decision will not affect your relationship with Northwestern University. You can leave the research at any time, and it will not be held against you.

### How will the researchers protect my information?

- We will use systematic protocols to collect your data. We also have a secured and private way for you to submit your data. This includes using a Virtual Private Network (VPN) connection for encryption and a SSH File Transfer Protocol (SFTP). SFTP allows secure transfer of private information, such as your name.
- We will store your data on secured, password-protected dataset servers behind passcodeprotected doors. Only our staff have access to your data with unique login info. Security access levels depends on the staff's roles for the project. For example, only staff who need to contact you will have access to your personal information. All the study staff have received training in ethnical research conduct.
- We will hide your name/address and will use a unique study ID to identify you.
- Our research team will handle all contact with you. You will not have contact with anybody who is not a trained member of this study.

#### Who will have access to the information collected during this research study?

We will limit the use and disclosure of your personal data to people who have a need to review this information. This includes research study records, but we cannot promise complete secrecy.

There are reasons why information about you may be used or seen by other people beyond the research team during or after this study. Examples include:

- University officials, government officials, study funders, auditors, and the Institutional Review Board may need access to the study information. This is to ensure that the study procedures are safe and appropriate.
- Collaborating researchers at other institutions who are involved with this study.
- The research team may give information to appropriate authorities for reasons of health and safety. This applies if you indicate that you plan to harm yourself or others, or for public health reasons.

We will not ask you about child abuse. But, if you tell us about child abuse or neglect, we may be required or permitted by law or policy to report to authorities.

Most tests done in research studies are only for research and have no clear meaning for your health.

If the research results have meaning for your health, the researchers will contact you to let you know what they have found.

### How might the information collected in this study be shared in the future?

We may share your de-identified data with the research community at large. This will help advancing science and health. We will remove or code any personal information that could identify you before sharing your data with other researchers. This ensures that no one can identify you from the information we share, which follows current scientific standards and known methods. However, we cannot guarantee complete anonymity.

### Will I be paid or given anything for taking part in this study?

You will receive \$100 as an online gift card upon completion of a focus group session for your participation in this study. There will not be any bonus payment. It will not cost you anything to be in this study.

#### Who can I talk to?

If you have questions, concerns, or complaints, you can contact the Principal Investigator Dr. Ricky Hill. Email: <u>ricky@northwestern.edu</u>; phone: 312-503-3610.

The Institutional Review Board ("IRB") has reviewed and approved this study. You may contact the IRB by phone at (312) 503-9338 or by email at <u>irb@northwestern.edu</u> if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

If you want a copy of this consent for your records, you can print it from the screen.

If you cannot print the consent and would like a copy for your records, contact the Principal Investigator with the contact information above.

If you wish to participate, please click the "I Agree" button and you will be taken to the brief demographic survey.

If you do not wish to participate in this study, please select "I Disagree" or select X in the corner of your browser.